CLINICAL TRIAL: NCT02433925
Title: Effects of Supplementation With Resveratrol on Inflammation and Oxidative Stress of Non-dialysis Chronic Kidney Disease Patients
Brief Title: Resveratrol's Effects on Inflammation and Oxidative Stress in Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DeniseMafra
Record Dates: First submitted 2015-02-19; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Renal Insufficiency
Keywords: resveratrol; oxidative stress; inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement B (Active Comparator): Administration of 500mg of trans-resveratrol per day, for 4 weeks
  Interventions: Dietary Supplement: Resveratrol
- Supplement A (Placebo Comparator): Administration of 500mg of placebo per day, for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol
  Other Names: trans-resveratrol
  Arms: Supplement B
Dietary Supplement: Placebo
  Arms: Supplement A

SUMMARY:
Inflammation and oxidative stress are common findings in patients with Chronic Kidney Disease (CKD) undergoing conservative treatment, in addition to being associated with atherosclerotic process, are related also to the progression of CKD. In this regard, resveratrol, a phenolic compound with recognized antioxidant and anti-inflammatory properties, can play an important role in the control of metabolic disorders associated with CKD, since it can modulate the mechanisms involved in inflammation and oxidative stress cycle. Resveratrol is capable of promoting the activation of the transcription-related factor-2 nuclear factor erythroid factor 2 (Nrf2) , a nuclear factor with anti-inflammatory properties, and SIRT-1, a protein also associated with the reduction of inflammation. These two factors, in their turn, are able to inhibit / antagonize the activity of the nuclear factor κB (NF-kB), a transcription factor that participates in the inflammatory response. Although it is a promising treatment, there are no studies evaluating the effects of resveratrol supplementation in patients with CKD. Thus, this study aims to evaluate the effects of resveratrol supplementation on inflammation and oxidative stress in patients undergoing conservative treatment of CKD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients in stages 3 or 4, undergoing conservative treatment

Exclusion Criteria:

* Patients with diabetes mellitus, AIDS, inflammatory or infectious diseases, pregnant women, smokers and those using antioxidant supplements

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Antioxidants and anti-inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers (Nrf2, GPx, HO-1)

SECONDARY OUTCOMES:
Inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory biomarkers (NFkB, IL-6, TNF-alfa)

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745